CLINICAL TRIAL: NCT04107571
Title: A Chinese Registry to Determine the Serumal Biomarkers for Prognosis of Adverse Events in Patients Undergoing Coronary Artery Bypass Grafting.
Brief Title: A Registry Study on Serumal Biomarkers About Adverse Events in Patients Undergoing Coronary Artery Bypass Grafting.
Acronym: ASBA-CABG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 20190924
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Surgery
Keywords: Coronary artery bypass graft; Biomarker; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If a blood specimen is obtained, it will be separated and stored at -80 ℃ as plasma, viable cells, and extracted DNA. If a saliva specimen is obtained, it is stored for DNA.
  If a tissue specimen is obtained, it will be cut into small pieces and stored at liquid nitrogen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort
  Interventions: Procedure: A type of operation for coranary heart disease patients.

INTERVENTIONS:
Procedure: A type of operation for coranary heart disease patients. — A type of operation for coranary heart disease patients.

SUMMARY:
This is a national registry study to determine the serumal biomarkers for prognosis of adverse events in patients undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject undergoing coronary artery bypass grafting;
2. Age is more than 18 and less than 80 years old;
3. Male and non pregnancy female;
4. Subject who understands study requirements and agrees to sign an informed consent from prior to study procedures.

Exclusion Criteria:

1. Pregnancy female;
2. Participate in other clinical trial in the last 1 month.
3. Subject who doesn't agree to sign an informed consent from prior to study procedures.
4. Subject undergoing repeat CABG, concomitant valve or other cardiac surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group consists of patients who underwent coronary artery bypass grafting in Beijing Anzhen Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
All-cause death and cardiac death | These data is collected during follow-up visit at in-hospital/1 year after discharge

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | These data is collected during follow-up visit at in-hospital/1 year after discharge
  A composite of death, myocardial infarction, stroke, heart failure, ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PHD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China